CLINICAL TRIAL: NCT00245388
Title: A Randomized, Double-Blind, Dose-Ranging, Placebo-Controlled Trial to Determine the Lipid-Lowering Efficacy and Safety of BMS-298585 Alone or in Combination With Pravastatin in Subjects With Mixed Dyslipidemia
Brief Title: Efficacy and Safety of BMS-298585 Alone or in Combination With Pravastatin in Subjects With Mixed Dyslipidemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-008
Record Dates: First submitted 2005-10-14; First posted 2005-10-28 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Dyslipidemia
Keywords: Mixed Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — muraglitazar

INTERVENTIONS:
Drug: Muraglitazar

SUMMARY:
This is a randomized, double-blind, dose-ranging, placebo-controlled trial to determine the lipid-lowering efficacy and safety of BMS-298585 (muraglitazar) alone in combination with pravastatin in subjects with mixed dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetics
* Serum TG >150 mg/dL and < or = 600 mg/dL
* Serum LDL-C >130 mg/dL

Exclusion Criteria:

* Type 1 or type 2 diabetics
* Fasting plasma glucose >126 mg/dL
* Treatment with lipid-lowering drugs, unless they can be withdrawn within the following time frame prior to the first qualifying lipid determination (Week 2):

  * Niacin or bile-acid binding agents and HMG CoA reductase inhibitors: 8 weeks
  * Fibrates: 8 weeks
  * Probucol: 1 year
* History of active liver disease and/or history of thiazolidinedione-related (troglitazone, rosiglitazone, or pioglitazone) liver abnormalities, hepatic dysfunction, or jaundice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2002-04; Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
To compare at a .05 level of significance, after 6 weeks of oral administration of double-blind treatment the percent change from baseline to average triglycerides (TG), week 5-6 between 5, 10 and 20 mg

SECONDARY OUTCOMES:
Percent changes from baseline to average at week 5-6 of total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-HDL-C, apolipoprotein A1 (ApoA1), and free fatty acid (FFA) levels

CONTACTS AND LOCATIONS:
Locations (54):
- United States (53):
  - Local Institution, Phoenix, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Irvine, California
  - Local Institution, Long Beach, California
  - Local Institution, Raleigh, California
  - Local Institution, Roseville, California
  - Local Institution, Sacramento, California
  - Local Institution, San Diego, California
  - Local Institution, Santa Ana, California
  - Local Institution, Longmont, Colorado
  - Local Institution, Clearwater, Florida
  - Local Institution, Cooper City, Florida
  - Local Institution, DeLand, Florida
  - Local Institution, Inverness, Florida
  - Local Institution, Longwood, Florida
  - Local Institution, Pembroke Pines, Florida
  - Local Institution, Sarasota, Florida
  - Local Institution, Stuart, Florida
  - Local Institution, Dunwoody, Georgia
  - Local Institution, Melbourne, Georgia
  - Local Institution, Peoria, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Iowa City, Iowa
  - Local Institution, Overland Park, Kansas
  - Local Institution, Wichita, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Marrero, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Bethesda, Maryland
  - Local Institution, Edina, Minnesota
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Toms River, New Jersey
  - Local Institution, Manlius, New York
  - Local Institution, Hickory, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Columbus, Ohio
  - Local Institution, Bend, Oregon
  - Local Institution, Hillsboro, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Sellersville, Pennsylvania
  - Local Institution, Warminster, Pennsylvania
  - Local Institution, Greer, South Carolina
  - Local Institution, Mt. Pleasant, South Carolina
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, San Angelo, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Olympia, Washington
  - Local Institution, Seattle, Washington
  - Local Institution, Yakima, Washington
- Local Institution, Ottawa, Ontario, Canada